CLINICAL TRIAL: NCT04249882
Title: A Novel Human Laboratory Model for Screening Medications for Alcohol Use Disorder
Brief Title: A Novel Human Lab Model for Screening AUD Medications
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Lara Ray, PhD, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-001735; R21AA027180 (NIH)
Record Dates: First submitted 2020-01-24; First posted 2020-01-31 (Actual); Results first posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-08

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol Use Disorder; Medications Development
MeSH Terms: conditions — Alcoholism | interventions — 5'-palmitoyl cytarabine; Naltrexone; Varenicline

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, 3-arm, parallel-group study of naltrexone (50 mg QD) and varenicline (1 mg BID).
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study team, medical personnel, and participants will be blind to drug condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo (Placebo Comparator): Matched to active medications
  Interventions: Drug: Placebo
- Varenicline (Active Comparator): 1 mg twice a day
  Interventions: Drug: Varenicline
- Naltrexone (Active Comparator): 50 mg once a day
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Placebo — Matched to active medication
  Other Names: PLAC
  Arms: Placebo
Drug: Naltrexone — 50 mg once a day
  Other Names: NTX
  Arms: Naltrexone
Drug: Varenicline — 1 mg twice a day
  Other Names: VAR; Chantix
  Arms: Varenicline

SUMMARY:
This study design consists of a randomized, double-blind, placebo-controlled, 3-arm, parallel-group study of naltrexone (50 mg QD) and varenicline (1 mg BID). A total of 108 men and women with current AUD (moderate or severe) and reporting intrinsic motivation to change their drinking, will be randomly assigned to receive naltrexone (50 mg QD), varenicline (1 mg BID) or matched placebo. Post-randomization, all participants will complete an alcohol cue-reactivity paradigm prior to the initial dose of study medication. After a week-long medication titration period, participants will be asked to complete a 7-day practice quit attempt, during which they will have daily virtual visits (phone and online) where they will report on their alcohol use. Additionally, a second cue-reactivity paradigm will be conducted 90 minutes following study drug administration on final day of the practice quit attempt (Day 14).

DETAILED DESCRIPTION:
Recruitment: Participants will be recruited from the community through online and newspaper advertisements. Campaigns in local buses and print publications (e.g., LA Weekly) will also be implemented. Targeted recruitment will also take place through a lab database of previous study participants who agreed to be contacted for future studies.

Telephone Screen: Individuals who call the lab (in response to flyers and advertisements) expressing interest in the study will receive detailed information about the study procedures, and if they remain interested they will complete a telephone screen performed by a trained research assistant for self-reported inclusion and exclusion criteria. Those who appear eligible will be invited to the laboratory for an initial in-person screening session.

Initial Screening: Prior to conducting any research related procedures, research staff will conduct the informed consent process, which details the procedures to take place during the screening visit. Informed consent will be a three-part process. First, participants will be asked to read and provide verbal consent for breathalyzer. If the breathalyzer is above 0.000, the visit will be stopped and the participant will not be compensated. The participant will be given an opportunity to reschedule the visit for another day. If the breathalyzer test is negative, the written informed consent form will be reviewed and signed by the participant and study staff outlining procedures for the initial screening visit. A second written consent form will be reviewed and signed in the presence of the study physician at the medical screening visit if the participant is found eligible to continue to that visit. At the initial screening visit, subjects will be asked to provide a urine sample to test for drugs of abuse and pregnancy (if female), and will complete a series of questionnaires and interviews (described in detail below) to determine initial eligibility. This visit will take approximately 1 hour. Following the initial in-person screening, the study coordinator will meet with the PI to determine if the participant is eligible to continue to the medical screening based on study inclusion/exclusion criteria.

Medical Screening: Those participants who appear to be eligible after the initial screening visit, will then be scheduled for a second screening visit. This visit will be conducted by the study physician and will start with a breathalyzer test. If the breathalyzer is above 0.000, the visit will be stopped and the participant will not be compensated. The participant will be given an opportunity to reschedule the visit for another day. If the breathalyzer test is negative, the physician will conduct the second written (experimental) consent; medical history interview and physical exam. In addition, a urine sample will be obtained for repeat drug screen and pregnancy tests. The participant will then be accompanied by research personnel to the CTRC for blood specimen collection including Comprehensive Metabolic Panel and Complete Blood Count to evaluate overall health; and EKG to screen for medical conditions that could make study participation medically unsafe. The study physician will review each participant's medical history, vital signs, weight, review of systems, and laboratory tests, including liver function tests (LFTs), drug screen, chemistry screen, and urine pregnancy screen to determine if it is medically safe for the participant to take the study medication. Any subject who is excluded from the study will be compensated for their time in the screening session and will be offered referrals for alcohol treatment in the community.

Randomization and Medication Titration: Participants who are eligible after the physical exam will be randomized to one of three treatment conditions (VAR, NTX, or PLA). Urn randomization will be used to balance the groups by gender, smoking status (as reported on question 1 of the Fagerstrom Test for Nicotine Dependence), and drinking status ('heavy' drinker defined as 28 or more drinks per week for males/14 or more drinks per week for females, or 'very heavy' drinker, defined as 35 or more drinks per week for males/28 or more drinks per week for females). The UCLA Research Pharmacy will manage the blind. The three treatment conditions will not be different in appearance or method of administration. All participants will undergo a week-long medication titration period prior to the onset of the practice quit attempt.

Practice-Quit Attempt: During the practice-quit attempt, participants will be instructed to abstain completely from drinking alcohol during a 7-day practice quit period. This period will begin on Day 8 of study medication dosing. During this period, participants will complete daily virtual visits to report on their drinking, mood and craving for alcohol during the previous day in a daily diary assessment (DDA).

Study Medication: On Day 1, participants will report to the laboratory to complete the alcohol cue-reactivity paradigm and receive their first medication dose under direct observation of study staff. They will receive a 7-day supply of study medication in blister packs with AM and PM dosing clearly distinguished for the titration procedure. After reaching full medication dose at the end of one week, participants will come to the laboratory on Day 8 to begin the practice quit attempt and to take AM dose of study medication daily in the lab under direct observation of study staff. Additionally, on the first day of the practice-quit attempt (Day 8), participants will receive a second 7-day supply of study medication. All study medication will be prepared by the UCLA Research Pharmacy and will be identically matched in appearance (opaque capsules with 50 mg of riboflavin to aid in medication compliance procedures) and the medication labels will not reveal the drug identity.

Alcohol Cue Reactivity Sessions (CR): Randomized participants will complete a cue-exposure paradigm at two time points during the study, once on Day 1 prior to ingesting the first dose of study medication, and again on Day 14, approximately 90 minutes after study drug administration. Alcohol cue exposure will follow well-established experimental procedures. Sessions will begin with a 3-minute relaxation period. Participants will then hold and smell a glass of water for 3 minutes to control for the effects of simple exposure to any potable liquid. Next, participants will hold and smell a glass of their preferred alcoholic beverage for 3 minutes. Order is not counterbalanced because of carryover effects that are known to occur. Participants (who are smokers) will be allowed a smoke break immediately prior to the CR assessment. After every 3 minutes of exposure, participants will rate their urge to drink on the Alcohol Urge Questionnaire (AUQ) and their mood on the Profile of Mood States (POMS). AUQ score (alcohol minus water) is the primary outcome for the CR.

Brief Counseling Session: All participants will meet with a trained study counselor briefly after the second cue exposure session on Day 14 to discuss their responses to the alcohol cues and discuss local treatment options. The counselor will begin by introducing him/herself and thanking the participant for his/her participation. He/she will continue by providing the participant with feedback on their responses on various individual difference measures (drinking patterns, severity of AUD diagnosis, family history, CIWA, depression, and other drug use). The counselor will probe for participants' attitudes towards these responses and diagnoses, and provide both informational and emotional support. Next, the counselor will go over the participant's history of alcohol treatment, in order to identify potential barriers to treatment access. He/she will discuss local treatment options with the participant, including the participant's primary care provider, self-help groups, and the UCLA Psychology Clinic. Lastly, the counselor will go over the "Rethinking Drinking" pamphlet with the participant, pointing out specific treatment options discussed in the session, and will address any questions or concerns.

ELIGIBILITY:
Inclusion Criteria:

1. Be between the ages of 21 and 65
2. Meet current (i.e., past 12-month) DSM-5 diagnostic criteria for AUD moderate or severe
3. Have intrinsic motivation to reduce or quit drinking (defined as self-reported intention to reduce or quit drinking within the next 6 months)
4. Report drinking at least 28 drinks per week if male (14 drinks per week if female) in the 28 days prior to the initial consent
5. Have reliable internet access

Exclusion Criteria:

1. Have a current (last 12 months) DSM-5 diagnosis of substance use disorder for any psychoactive substances other than alcohol and nicotine
2. Have a lifetime DSM-5 diagnosis of schizophrenia, bipolar disorder, or any psychotic disorder
3. Have a positive urine screen for drugs other than cannabis
4. Have clinically significant alcohol withdrawal symptoms as indicated by a score ≥ 10 on the Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-R)
5. Have an intense fear of needles or have had any adverse reactions to needle puncture
6. Be pregnant, nursing, or planning to become pregnant while taking part in the study; and must agree to one of the following methods of birth control (if female), unless she or partner are surgically sterile:

   * Oral contraceptives
   * Contraceptive sponge
   * Patch
   * Double barrier
   * Intrauterine contraceptive device
   * Etonogestrel implant
   * Medroxyprogesterone acetate contraceptive injection
   * Complete abstinence from sexual intercourse
   * Hormonal vaginal contraceptive ring
7. Have a medical condition that may interfere with safe study participation (e.g., unstable cardiac, renal, or liver disease, uncontrolled hypertension or diabetes)
8. Be currently taking any psychotropic medications that, in the opinion of the investigators, compromises participant safety
9. Be currently taking or have had previous experience with either naltrexone or varenicline
10. Have any other circumstances that, in the opinion of the investigators, compromises participant safety

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lara Ray, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Addictions Lab, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baskerville WA, Grodin EN, Meredith LR, Ray LA. Interplay between alcohol cues and mood states during early abstinence: A daily diary study. Exp Clin Psychopharmacol. 2025 Jun;33(3):260-268. doi: 10.1037/pha0000770. Epub 2025 Mar 13. PMID 40080609
- [Derived] Ho D, Towns B, Grodin EN, Ray LA. A novel human laboratory model for screening medications for alcohol use disorder. Trials. 2020 Nov 23;21(1):947. doi: 10.1186/s13063-020-04842-w. PMID 33225963

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via online and print advertisements, local bus campaigns, and targeted recruitment through a laboratory database of previous study participants who agreed to be contacted for further studies.
Pre-assignment Details: A stratified randomization list was developed by a statistician and was based on gender, smoking status (as reported on the Fagerstrom Test for Nicotine Dependence (FTND; (Heatherton et al. 1991)), and drinking status ('heavy' drinker defined as ≥ 14 for males/ ≥7 for females, or 'very heavy' drinker defined as ≥35 for males/≥ 28 for females).
Period: Overall Study
Arm/Group | Placebo | Varenicline | Naltrexone
Started | 19 | 19 | 15
Completed | 17 | 17 | 14
Not Completed | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Varenicline | Naltrexone | Total
Number analyzed (Participants) | 19 | 19 | 15 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.47 (11.91) | 41.84 (13.04) | 42.40 (11.19) | 41.87 (11.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 7 | 26
  Male | 10 | 9 | 8 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 3 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 5 | 5 | 4 | 14
  White | 7 | 9 | 7 | 23
  More than one race | 4 | 3 | 2 | 9
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 15 | 53
Last 30 Days Drinks Per Drinking Day [Mean (Standard Deviation); unit: number of drinks per drinking day] | 5.46 (2.39) | 5.84 (3.68) | 5.89 (3.48) | 5.73 (3.18)
Past Month Percent Day Abstinent [Mean (Standard Deviation); unit: percent days abstinent] | 25.79 (21.16) | 28.78 (24.92) | 25.56 (23.12) | 28 (23.19)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Days Abstinent
Description: The percentage of days abstinent from alcohol is determined using the Timeline Follow Back (TLFB). The TLFB was administered to assess quantity and frequency of alcohol use each day during the practice quit period (Day 8 - Day 14). Information obtained in this interview was recorded on the TLFB Calendar and transcribed to a database. The primary outcome variable was calculated as the percent of days participants were abstinent during the practice quit period.
Time Frame: 6 days
Measure: Least Squares Mean (Standard Error); unit: percent days
Arm/Group | Placebo | Varenicline | Naltrexone
Number analyzed (Participants) | 17 | 17 | 14
percent days | 80.59 (6.67) | 75.62 (6.87) | 77.59 (7.31)

2. Primary Outcome: # of Drinks Per Drinking Day
Description: The drinks per drinking day outcome is determined using the the Timeline Follow Back (TLFB). The TLFB was administered to assess quantity and frequency of alcohol use each day during the practice quit period (Day 8 - Day 14). Information obtained in this interview was recorded on the TLFB Calendar and transcribed to a database. The primary outcome variable was calculated as the number of drinks per drinking day during the practice quit period.
Time Frame: 6 days
Measure: Least Squares Mean (Standard Error); unit: number of drinks per drinking day
Arm/Group | Placebo | Varenicline | Naltrexone
Number analyzed (Participants) | 17 | 17 | 14
number of drinks per drinking day | 1.66 (0.63) | 2.19 (0.65) | 2.73 (0.69)

3. Primary Outcome: Cue-induced Craving
Description: Randomized participants completed a cue-exposure paradigm at two time points during the study, once on Day 1 prior to ingesting the first does of study medication, and again on Day 14. After every 3 minutes of exposure (water and alcohol), participants rated their urge to drink on the Alcohol Urge Questionnaire (AUQ). The AUQ is comprised of eight items rated on a 7-point Likert scale with items related to the subjective experience of alcohol craving, with higher total scores indicating higher craving and a minimum score of 8 and maximum score of 56. Alcohol urge questionnaire score (alcohol minus water) is the primary outcome for the cue-reactivity paradigm. The investigators are primarily interested in the difference in craving from post-treatment (day 14) to pre-treatment (randomization/day 1).
Time Frame: Cue reactivity paradigm takes place on Day 1 and on Day 14. Craving is measured 3 min after each cue exposure
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Varenicline | Naltrexone
Number analyzed (Participants) | 19 | 19 | 15
units on a scale | -0.11 (0.35) | 0.31 (0.33) | -0.32 (0.37)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each participant between randomization to Day 14 (final day of study).
Description: Adverse event data was collected on a daily basis during the practice quit using the 24 items form the side effects checklist (SAFTEE) ) (Jacobson et al. 1986; Levine and Schooler 1986).
Arm/Group | Placebo | Varenicline | Naltrexone
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/15
Other Adverse Events (participants affected / at risk) | 15/19 | 13/19 | 14/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=19) | Varenicline (N=19) | Naltrexone (N=15)
Abdominal Pain or Cramps (Gastrointestinal disorders) | 3 | 4 | 4
Yellow Eyes (Eye disorders) | 2 | 1 | 1
Nausea or Vomiting (Gastrointestinal disorders) | 1 | 5 | 3
Irritability or Anger (Psychiatric disorders) | 5 | 6 | 10
Increased Desire for Sex (Reproductive system and breast disorders) | 6 | 5 | 5
Nervousness (Psychiatric disorders) | 5 | 5 | 7
Ringing in the Ears (Ear and labyrinth disorders) | 0 | 2 | 3
Decrease in Appetite (General disorders) | 2 | 4 | 4
Depression (Psychiatric disorders) | 4 | 4 | 3
Fatigue (General disorders) | 8 | 8 | 8
Difficulty in Staying Awake (General disorders) | 4 | 3 | 4
Increase in Appetite (Metabolism and nutrition disorders) | 4 | 4 | 6
Blurred Vision (Eye disorders) | 1 | 0 | 2
Drowsiness (General disorders) | 3 | 10 | 3
Headache (General disorders) | 3 | 6 | 5
Night Sweats (General disorders) | 2 | 2 | 4
Mental Confusion (Psychiatric disorders) | 2 | 2 | 2
Anxiety (Psychiatric disorders) | 5 | 7 | 9
Joint or Muscle Pain (General disorders) | 1 | 4 | 8
Dizziness (General disorders) | 1 | 3 | 3
Sexual Problems (Reproductive system and breast disorders) | 0 | 1 | 2
Difficulty Sleeping (General disorders) | 6 | 6 | 8
Fever or Chills (General disorders) | 0 | 1 | 1
Decreased Desire for Sex (Reproductive system and breast disorders) | 1 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT04249882/Prot_SAP_001.pdf